CLINICAL TRIAL: NCT05343156
Title: Efficacy and Safety of Dexamethasone Nanoparticles Eye Drops in Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oculis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DX211
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DexNP Eye Drop (Experimental): The study eye received 1 DexNP eye drop 3 times a day (every 8 hours) for 12 weeks.
  Interventions: Drug: Dexamethasone nanoparticles eye drops
- Vehicle Eye Drop (Placebo Comparator): The study eye received 1 vehicle eye drop 3 times a day (every 8 hours) for 12 weeks.
  Interventions: Drug: Dexamethasone nanoparticles eye drops

INTERVENTIONS:
Drug: Dexamethasone nanoparticles eye drops — DexNP 15 mg/mL eye drops 3 times a day (every 8 hours) for 12 weeks

SUMMARY:
Anti-inflammatory or anti-angiogenic drugs play an ever- increasing role in the treatment of diabetic macular edema (DME). The drug delivery systems, such as injections of corticosteroid and or vascular endothelial growth factor (VEGF) antibodies into the vitreous cavity or slow release drug capsules surgically implanted in the eyes run the risk of surgical complications including infections, hemorrhages and cataracts and place a huge demand on eye care resources significantly increase the risk of cardiovascular events and death.

A non-invasive drug delivery platform with steroid eye drops, reaching the back of the eye to treat DME and other retinal diseases would circumvent most of these problems.

A novel drug delivery platform is required for ocular therapy. Oculis ehf. has developed a drug delivery platform, which is based on cyclodextrin nanoparticles that dissolve in the tear fluid to form water-soluble drug/cyclodextrin complex nanoparticles. Animal and initial clinical testing has shown the potential for this technology to increase the drug concentration in the eye tissues including the retina and therefore treat retinal diseases like DME.

ELIGIBILITY:
Key Inclusion Criteria:

1. Had DME of less than 3 years duration since diagnosis with presence of intraretinal and/or subretinal fluid in the study eye, with CMT of ≥ 310 µm by SD-OCT at baseline (Visit 2) (as measured by the Investigator).
2. Had definite retinal thickening in the study eye due to DME involving the central macula based on the Investigator's clinical evaluation and by SD-OCT;

   ...

Key Exclusion Criteria:

1. Had macular edema considered to be due to a cause other than DME;
2. Had a decrease in BCVA due to causes other than DME (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, previous vitreoretinal surgery, central serous retinopathy, non-retinal condition, substantial cataract, macular ischemia) that is likely to be decreasing BCVA by 3 lines or more (i.e., cataract would be reducing acuity to 20/40 or worse if eye was otherwise normal).

   ...

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Larsen, MD, Study Director — Glostrup University Hospital, Copenhagen
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Denmark

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DexNP Eye Drop | Vehicle Eye Drop
Started | 99 | 45
Completed | 91 | 42
Not Completed | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DexNP Eye Drop | Vehicle Eye Drop | Total
Number analyzed (Participants) | 99 | 45 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (9.5) | 66.1 (9.92) | 64.4 (9.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 17 | 52
  Male | 64 | 28 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 98 | 45 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Early Treatment of Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA)
Description: The primary efficacy endpoint was summarized by treatment group using descriptive statistics, including 70%, 90% and 95% confidence intervals (CIs). Change from baseline to Week 12 is also summarised by treatment group.
  The primary analysis of the primary endpoint employed a linear model with change from baseline ETDRS BCVA letters as the response, baseline ETDRS BCVA letters as a covariate, and treatment as a main effect factor, using the ITT population and with multiple imputation pattern mixture model techniques used to impute missing data.
Time Frame: Baseline & Week 12
Population: Change from baseline to week 12 in Study Eye ETDRS BCVA Letters using Multiple Imputation (Intent-to-Treat Population)
Measure: Least Squares Mean (70% Confidence Interval); unit: ETDRS BCVA Letters
Arm/Group | DexNP Eye Drop | Vehicle Eye Drop
Number analyzed (Participants) | 99 | 45
ETDRS BCVA Letters | 2.62 [1.831 to 3.403] | 1.04 [-0.115 to 2.189]

ADVERSE EVENTS:
Time Frame: Subjects were monitored for safety on all study visits. Assessment of AEs, including definition of seriousness, severity and causality was performed at each visit : day 1 (visit 2), week 2 (visit 3), week 4 (visit 4), week 8 (visit 5) , week 12 (visit 6) and week 16 (visit 7)
Arm/Group | DexNP Eye Drop | Vehicle Eye Drop
All-Cause Mortality (participants affected / at risk) | 2/99 | 0/45
Serious Adverse Events (participants affected / at risk) | 11/99 | 1/45
Other Adverse Events (participants affected / at risk) | 32/99 | 9/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DexNP Eye Drop (N=99) | Vehicle Eye Drop (N=45)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Endocrine disorders) | 1 (2) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
diabetic ulcer (Endocrine disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DexNP Eye Drop (N=99) | Vehicle Eye Drop (N=45)
Intraocular pressure increased (Investigations) | 21 (23) | 0 (0)
Blood glucose fluctuation (Investigations) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 3 (3) | 0 (0)
Ocular hypertension (Eye disorders) | 3 (3) | 0 (0)
Cataract subcapscular (Eye disorders) | 1 (1) | 1 (1)
conjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinal edema (Eye disorders) | 1 (1) | 0 (0)
erythema of eyelid (Eye disorders) | 1 (1) | 1 (1)
eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
glaucoma (Eye disorders) | 1 (1) | 0 (0)
noninfective conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperemia (Eye disorders) | 1 (1) | 1 (1)
photophobia (Eye disorders) | 1 (1) | 0 (0)
posterior capsule opacification (Eye disorders) | 1 (1) | 1 (1)
conjunctival hyperemia (Eye disorders) | 0 (0) | 1 (1)
conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
corneal edema (Eye disorders) | 0 (0) | 1 (1)
eye infection bacterial (Eye disorders) | 0 (0) | 1 (1)
eye pruritus (Eye disorders) | 0 (0) | 1 (1)
foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1)
keratopathy (Eye disorders) | 0 (0) | 1 (1)
retinal pigment epitheliopathy (Eye disorders) | 0 (0) | 1 (1)
dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
eye infection bacterial (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees not to publish/present the results until such time as the aggregate study results are published. After such time, Investigator may publish the results in accordance with the following: Investigator shall submit to Sponsor any such proposed publication/presentation resulting from or relating to the Study at least 60 days prior to the submission for publication. Sponsor may require the delay of publication/presentation for an additional period of time not to exceed 120 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT05343156/Prot_SAP_000.pdf